CLINICAL TRIAL: NCT00146003
Title: Investigator-Initiated Trial of Efalizumab for Atopic Dermatitis: A Proof of Concept Study in Adults
Brief Title: Efalizumab for Eczema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: Genentech, Inc. (Industry)
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5163
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2008-08-07 (Estimated); Status verified 2008-08

CONDITIONS: Dermatitis, Atopic
Keywords: eczema; atopic dermatitis; efalizumab
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Efalizumab treatment

SUMMARY:
The purpose of this study is to demonstrate a measurable improvement on a validated scale in a small population of adult patients with atopic dermatitis (eczema).

DETAILED DESCRIPTION:
The study involves administration of efalizumab (previously approved for psoriasis) to ten adult patients with atopic dermatitis. Biologic plausibility rests on similarities in pathophysiology of the two conditions. The drug (efalizumab) will be administered according to the dosing approved for plaque psoriasis for a period of 24 weeks. The subjects will self-administer efalizumab weekly and measurements will be performed on a monthly basis. Efalizumab is not being compared to placebo or other drugs.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or older) with atopic dermatitis with 5% or more body surface area involvement
* Investigator Global Assessment (IGA) score of "moderate" or worse
* In general good health with well-controlled medical problems
* Ability to provide written informed consent and comply with study assessments for the full duration of the study.
* If a female of childbearing potential, a negative pregnancy test and commitment to the use of two forms of effective contraception (birth control) for the duration of the study are necessary.
* If a non-sterile male, commitment to the use of two forms of effective contraception (birth control) for the duration of the study is necessary.
* Normal platelet count

Exclusion Criteria:

* Patients with known hypersensitivity to efalizumab or any of its components
* Pregnancy or lactation
* Patients receiving immunosuppressive agents
* Prior enrollment in the study
* Participation in another simultaneous medical investigation or trial
* IGA score of "mild," "almost clear" or "clear"
* Systemic therapy for atopic dermatitis, phototherapy or topical therapy (other than moisturizer) within 1 week
* Medical condition which would make use of efalizumab unsafe; would limit compliance with study requirements; or would limit accurate assessment of efficacy.
* Ongoing, active, serious infection
* History of malignancy (except excised basal or squamous cell carcinoma of the skin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2005-03; Study Completion 2007-12

PRIMARY OUTCOMES:
Percent of subjects achieving "clear" to "almost clear" on the Investigator Global Assessment [IGA] (success is achieved if 2 of 10 patients achieve "clear" or "almost clear" at any point in the study)

SECONDARY OUTCOMES:
Percent of subjects achieving "mild," "almost clear," or "clear" on the IGA
Percent improvement from baseline on the EASI (eczema area and severity index)
Photography (quarter-body views, front and back)
Pruritus improvement from baseline (rated on a scale of 1 to 10)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Magliocco, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- UMDNJ Psoriasis Center of Excellence, New Brunswick, New Jersey, United States